CLINICAL TRIAL: NCT03226171
Title: Dose Adjustment Trial of SK-1403 in Hemodialysis Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJ1002
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-adjusted SK-1403 (Experimental)
  Interventions: Drug: Dose-adjusted SK-1403

INTERVENTIONS:
Drug: Dose-adjusted SK-1403 — SK-1403 is to be administered to patients for the whole treatment periods (52 weeks), with individual dose adjustment

SUMMARY:
This study is conducted to assess the efficacy and safety of SK-1403 in Hemodialysis Patients with Secondary Hyperparathyroidism. In the first treatment period, the efficacy of SK-1403 is assessed after 18 weeks of treatment with SK-1403 individually dose-adjusted . Safety is also assessed during this period. Patients who completed the first treatment period proceed to the second treatment period and receive the treatment with SK-1403 for 34 weeks. Efficacy and safety of SK-1403 are also assessed during this period.

ELIGIBILITY:
Inclusion Criteria:

* Average serum PTH>240 pg/mL during 2 weeks at the screening
* Serum corrected Ca≧8.4 mg/dL at the screening
* Stable chronic kidney disease patients who undergo hemodialysis or hemodialysis filtration

Exclusion Criteria:

* Primary hyperparathyroidism
* Severe liver disease
* Severe Cardiac disease
* History or family history of Long QT syndrome
* Malignant tumor
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* A history of severe drug allergy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients who achieved serum PTH between 60 pg/mL and 240 pg/mL, inclusive | 18 weeks
  Assessed by laboratory test value

SECONDARY OUTCOMES:
Rate of patients who achieved ≥ 30% or 50% reduction in serum PTH from baseline, respectively | 18 weeks
  Assessed by laboratory test value
Measured values and Changes from baseline in serum PTH, Ca, P, and serum Ca x P product | 52 weeks
  Assessed by laboratory test value

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan